CLINICAL TRIAL: NCT04536870
Title: STAREE-HEART Sub-study Clinical Trial
Brief Title: Statins in Reducing Events in the Elderly (STAREE) Heart Sub-study
Acronym: STAREE-HEART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Curtin University (Other)
Responsible Party: Principal Investigator, Ingrid Hopper, Principal Investigator, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APP1165440
Record Dates: First submitted 2020-08-25; First posted 2020-09-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Atrial Fibrillation; Healthy Ageing; Hypercholesterolemia; Myocardial Dysfunction
Keywords: Statin; Atorvastatin; STAREE; Echocardiography; Atrial fibrillation screening; Global longitudinal strain; Single time point screening; Elderly
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation; Hypercholesterolemia | interventions — Echocardiography; Global Longitudinal Strain; Electrocardiography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STAREE Statin group (Experimental): Participants in STAREE trial randomised to statin
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: ECG screening
- STAREE Placebo group (Experimental): Participants in STAREE trial randomised to placebo
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: ECG screening

INTERVENTIONS:
Diagnostic Test: Echocardiography — Ultrasound of heart
  Other Names: Global longitudinal strain
Diagnostic Test: ECG screening — Single lead ECG screening twice daily for two weeks
  Other Names: Alivecor
Diagnostic Test: ECG Screening — 12-lead ECG screening
  Other Names: 12-lead ECG

SUMMARY:
The STAREE-HEART sub-study will examine the effect of statin treatment over a 3-year period compared with placebo on markers of cardiac ageing (myocardial dysfunction). This will include determining global longitudinal strain with transthoracic echocardiography, atrial fibrillation with home measures twice daily for two weeks and changes in biomarkers.

DETAILED DESCRIPTION:
STAREE-HEART is an ancillary study nested in the Statins in Reducing Events in the Elderly (STAREE) double-blind randomised placebo-controlled trial. STAREE is investigating whether statins can prolong good health and maintain independence amongst older people and is enrolling men and women 70 years of age and over who are free from cardiovascular disease, diabetes and dementia. STAREE-HEART will recruit a subset of STAREE participants before they are randomised to STAREE study drug. STAREE-HEART will involve an additional suite of cardiac assessments in these participants and will provide detailed information about the clinical effect of statins on myocardial function.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥70 years living independently in the community who are participants in the STAREE RCT and eligible for randomisation to study medication.
* Willing and able to provide informed consent and accept the STAREE-HEART study requirements, including attendance for an echocardiogram and undertaking home monitoring via ECG.

Exclusion Criteria:

* Known atrial fibrillation or atrial flutter.
* Participants who do not wish to be informed of an abnormality under any circumstances, regardless of severity, will not be enrolled in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 369 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Global longitudinal strain (GLS) measured via transthoracic echocardiography. | 3 years
  Change in global longitudinal strain.

SECONDARY OUTCOMES:
Atrial fibrillation (AF) measured via single lead handheld ECG recordings. | 3 years
  Development of new AF.
Wavelet analysis via 12-lead ECG with Energy Waveform displays. | 3 years
  Increases detection of Heart Failure (HF).

OTHER OUTCOMES:
Atrial strain | Baseline to 3 year
  On echocardiography
N- Terminal-pro-Brain Natriuretic Peptide (NT pro BNP) | Baseline to 3 year
  Predictor of heart failure
Vascular Endothelial Growth Factor (VEG-F) | Baseline to 3 year
  Endothelial marker
Intercellular Adhesion Molecule 1 (ICAM-1) | Baseline to 3 year
  Endothelial marker
C-reactive protein | Baseline to 3 year
  Inflammatory biomarker
Interleukin-6 | Baseline to 3 year
  Inflammatory biomarker
Tumour Necrosis Factor alpha (TNF alpha) | Baseline to 3 year
  Inflammatory biomarker
Matrix metalloproteinase-9 (MMP-9) | Baseline to 3 year
  Fibrosis marker
Tumour-derived protein tissue inhibitor of metalloproteinases-1 (TIMP-1) | Baseline to 3 year
  Fibrosis marker
C-telopeptide of type I collagen (CTX I) | Baseline to 3 year
  Fibrosis marker
Procollagen III N-terminal propeptide (PIIINP). | Baseline to 3 year
  Fibrosis marker

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Hopper, Principal Investigator — Monash University; Sophia Zoungas, MBBS PhD FRACP, Study Chair — Monash University
Locations (2):
- Australia (2):
  - Monash University; School of Public Health and Preventative Medicine: STAREE trial, Melbourne, Victoria
  - Curtin University, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No
On completion of the trial, and after publication of the primary and secondary outcomes of the study, requests for access to de-identified data (to be provided through a secure online environment) may be submitted to the researchers located at the School of Public Health and Preventive Medicine, Monash University, Melbourne, Australia

REFERENCES:
- [Derived] Hopper I, Marwick TH, Wolfe R, Amerena J, Curtis AJ, Freedman B, Green DJ, Kaye D, Kolomoisky A, McNeil JJ, Nelson MR, Reid CM, Spark S, Tonkin AM, Wang BH, Zhou Z, Zoungas S. STAREE-HEART: A randomized placebo-controlled trial of atorvastatin effects on a marker of cardiac aging in older individuals without prior cardiovascular disease events: Protocol and baseline description of participants. Am Heart J. 2025 Dec;290:140-152. doi: 10.1016/j.ahj.2025.06.004. Epub 2025 Jun 12. PMID 40516583